CLINICAL TRIAL: NCT05281744
Title: Collaborative Care Coordination Program for Alzheimer's Disease and Related Dementias (Co-CARE-AD)
Brief Title: Collaborative Care Coordination Program for Alzheimer's Disease and Related Dementias
Acronym: Co-CARE-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Tufts Health Plan (Unknown); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Xiaojuan Li, Instructor in Population Medicine, Harvard Medical School and Harvard Pilgrim Health Care Institute, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AH000843; 5U54AG063546-03 (NIH)
Record Dates: First submitted 2022-02-25; First posted 2022-03-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2024-10

CONDITIONS: Alzheimer's Disease and Related Dementias (ADRD)
Keywords: dementia; informal caregiver; care consultation; care coordination
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dementia Care Consultation program (Experimental): The Dementia Care Consultation program provides an in-depth, personalized service for individuals and families facing ADRD.
  Interventions: Behavioral: Dementia Care Consultation program
- Routine Care (No Intervention): Members randomized into the control group will receive routine care.

INTERVENTIONS:
Behavioral: Dementia Care Consultation program — The Dementia Care Consultation program uses a telephone-based intervention to provide an in-depth, personalized service for individuals living with ADRD and their care partners. It consists of comprehensive needs assessments, creation and implementation of personalized care plans, monitoring and revising care plans, disease education and support coaching, referrals to community-based organizations for service and support, and access to assistance.
  Arms: Dementia Care Consultation program

SUMMARY:
This is a randomized, pragmatic clinical trial to evaluate the effectiveness of a collaborative care-coordination program embedded in a health plan for people living with Alzheimer's disease and related dementias (ADRD) and their care partners versus usual care. The study population will include community-dwelling Medicare Advantage members living with ADRD and their care partners. Outcomes will be healthcare utilization outcomes of individuals with ADRD and include emergency department visits, outpatient visits, avoidable emergency department visits, and admission to long-term care facilities.

ELIGIBILITY:
Community-dwelling Tufts Health Plan Medicare Advantage members with ADRD and their caregivers will be selected to participate in the trial based on the following inclusion/exclusion criteria:

Inclusion Criteria (for members with ADRD)

* Member of Tufts Health Plan Medicare Advantage plan
* Medical and pharmacy insurance coverage in at least the prior 12 months
* Have ≥1 ICD-10-CM diagnosis code for ADRD or dispensing for pharmacological treatment for ADRD in the prior 12 months

Exclusion Criteria (for members with ADRD):

* Reside in a nursing home or skilled nursing facility
* Enrolled in a hospice program
* Receiving or have received the Dementia Care Consultation program as part of the existing program at the time of enrollment

Inclusion Criteria (for caregivers)

* Age 18 years or older
* Assume primary responsibility for members

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2160 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
All-cause emergency department visits | by 12 months
  Number of all-cause emergency department visits per member living with ADRD over the 12-month follow-up period.
All-cause emergency department visits | by 6 months
  Number of all-cause emergency department visits per member living with ADRD over the 6-month follow-up period.

SECONDARY OUTCOMES:
Outpatient visits | by 12 months
  Number of outpatient visits per member living with ADRD over the 12-month follow-up period.
Outpatient visits | by 6 months
  Number of outpatient visits per member living with ADRD over the 6-month follow-up period.
Avoidable emergency department visits | by 12 months
  Number avoidable emergency department visits (defined using the validated New York University ED visit algorithm) per member living with ADRD over the 12-month follow-up period.
Avoidable emergency department visits | by 6 months
  Number avoidable emergency department visits (defined using the validated New York University ED visit algorithm) per member living with ADRD over the 6-month follow-up period.
Admission to long-term care facilities | by 12 months
  Number of members living with ADRD with the first admission to long-term care facilities over the 12-month follow-up period.
Admission to long-term care facilities | by 6 months
  Number of members living with ADRD with the first admission to long-term care facilities over the 6-month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojuan Li, PhD MSPH, Principal Investigator — Harvard Pilgrim Health Care Institute; Richard Platt, MD MS, Principal Investigator — Harvard Pilgrim Health Care Institute
Locations (1):
- Tufts Health Plan, Watertown, Massachusetts, United States